CLINICAL TRIAL: NCT02767323
Title: Using fMRI-guided TMS to Increase Central Executive Function in Older Adults
Brief Title: Using TMS to Increase Executive Function in Older Adults
Acronym: WMTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00065334; 1R01AG050618-01 (NIH)
Record Dates: First submitted 2016-05-05; First posted 2016-05-10 (Estimated); Results first posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Aging

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Active or Sham rTMS over the DLPFC (Aim1a) (Experimental): excitatory rTMS applied over the DLPFC (fMRI-guided). Active and Sham rTMS will be tested in a within subject design
  Interventions: Device: rTMS; Device: Sham rTMS
- Active or Sham rTMS over the Parietal cortex (Aim1b) (Experimental): excitatory rTMS applied over the parietal cortex (fMRI-guided). Active and Sham rTMS will be tested in a within subject design
  Interventions: Device: rTMS; Device: Sham rTMS
- Active or Sham rTMS over the DLPFC and the Parietal cortex (Aim1c) (Experimental): excitatory rTMS applied over the DLPFC and the parietal cortex (fMRI-guided). Active and Sham rTMS will be tested in a within subject design
  Interventions: Device: rTMS; Device: Sham rTMS

INTERVENTIONS:
Device: rTMS — excitatory 5Hz rTMS will be used
Device: Sham rTMS — an electrical sham coil reproducing the same clicking sound and tactile sensation than the active rTMS will be used

SUMMARY:
Cognitive decline and dementia have become important public health issues in our time as medical science has increased lifespan and our society becomes progressively older. A great deal of the cognitive decline due to aging can be explained by decline in working memory (WM), a mental function central to cognition in which aging deficits appear almost universally. Attempts to use WM training to increase WM ability in older adults has had some success, but the transfer of performance enhancements caused by this training to other cognitive skills is controversial. Another intervention that shows much promise is noninvasive stimulation of cerebral cortex using transcranial magnetic stimulation (TMS), which has been shown to increase performance in many cognitive tasks.

Here, the investigator proposes to use fMRI-guided rTMS to enhance working memory performance. This will be achieved through three Aims. In the first, registered on this record, the investigator will stimulate both old and young healthy adults while they perform the WM task that will engage the frontoparietal network. To define the optimal rTMS target, rTMS will be applied over the dorsolateral prefrontal cortex (DLPFC: Aim 1a); or over the parietal cortex (PC: Aim 1b). These regions are involved not only in the maintenance of items in WM, but also in their manipulation, therefore applying rTMS over these areas should create WM performance enhancements that will be long-lasting. In Aim 1c, a direct within-subject comparison of these 2 targeted sites is performed.

In the second and third Aims, older adults will receive active or sham rTMS over the optimal target (defined in Arm 1) during two weeks of daily sessions while they perform the WM tasks. In the second Aim, the investigator hopes to demonstrate that the cumulative effect of multiple TMS sessions, in tandem with the synergistic effects of simultaneous TMS + WM training, create WM performance enhancements greater than those found with WM training alone, whose effects are long-lasting, continuing a month following the course of TMS sessions. In the third, the investigator will investigate whether the WM enhancements generated by the two weeks of TMS sessions will generalize to other cognitive tasks. The success of these 3 Aims will provide proof in principle for long-lasting, transferable effects of TMS in remediating WM and more general cognitive deficits due to aging, and point to a possible non-invasive brain stimulation therapy for cognitive decline in healthy aging and in dementia. This record is a reflection of Aim1, Aim 2 and 3 will be registered separately.

ELIGIBILITY:
Inclusion Criteria:

* Age Restrictions: Young Group (from 18 to 35 years old), Elderly Group (from 60 to 80 years old).
* Use of effective method of birth control for women of childbearing capacity.
* Willing to provide informed consent.

Exclusion Criteria:

* Current or recent (within the past 6 months) history of substance abuse or dependence.
* Current serious medical illness.
* History of seizure, epilepsy, stroke, brain surgery, head injury, cranial metal implants, known structural brain lesion, devices that may be affected by rTMS or MRI (pacemaker, medication pump, cochlear implant, implanted brain stimulator)
* Inability or unwilling to give informed consent.
* Diagnosed any Axis I DSM-IV disorder (MINI, DSM-IV).
* For subjects age > 59 years, a total scaled score < 8 on the Dementia Rating Scale-2.
* Clinically defined neurological disorder.
* Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure, or currently taking medication that lowers the seizure threshold.
* Claustrophobia (MRI scanner).
* Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Appelbaum, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Crowell CA, Davis SW, Beynel L, Deng L, Lakhlani D, Hilbig SA, Palmer H, Brito A, Peterchev AV, Luber B, Lisanby SH, Appelbaum LG, Cabeza R. Older adults benefit from more widespread brain network integration during working memory. Neuroimage. 2020 Sep;218:116959. doi: 10.1016/j.neuroimage.2020.116959. Epub 2020 May 20. PMID 32442638

RESULTS

PARTICIPANT FLOW:
Groups:
- Active or Sham rTMS Over the DLPFC (Aim1a): excitatory rTMS applied over the DLPFC (fMRI-guided)
  rTMS: excitatory 5Hz rTMS will be used Active and Sham rTMS will be tested in a within subject design
- Active or Sham rTMS Over the Parietal Cortex (Aim1b): excitatory rTMS applied over the parietal cortex (fMRI-guided)
  rTMS: excitatory 5Hz rTMS will be used Active and Sham rTMS will be tested in a within subject design
- Active or Sham rTMS Over the DLPFC and the Parietal Cortex (Aim 1c): excitatory rTMS applied over the the DLPFC and the parietal cortex (fMRI-guided)
  rTMS: excitatory 5Hz rTMS will be used. Active and Sham rTMS will be tested in a within subject design
- Active/Sham rTMS Over DLPFC (Aim1a), Then Active/Sham rTMS Over DLPFC and Parietal Cortex (Aim1c): excitatory rTMS applied over the DLPFC (fMRI-guided) and the Parietal cortex
  rTMS: excitatory 5Hz rTMS will be used Active and Sham rTMS will be tested in a within subject design
Period: Overall Study
Arm/Group | Active or Sham rTMS Over the DLPFC (Aim1a) | Active or Sham rTMS Over the Parietal Cortex (Aim1b) | Active or Sham rTMS Over the DLPFC and the Parietal Cortex (Aim 1c) | Active/Sham rTMS Over DLPFC (Aim1a), Then Active/Sham rTMS Over DLPFC and Parietal Cortex (Aim1c)
Started | 83 | 42 | 58 | 1
Completed | 49 | 17 | 28 | 1
Not Completed | 34 | 25 | 30 | 0
Not completed — Withdrawal by Subject | 17 | 5 | 13 | 0
Not completed — Contraindication, moving during the scan, low behavior, or Covid-19 | 17 | 20 | 17 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active or Sham rTMS Over the DLPFC (Aim1a): excitatory rTMS applied over the DLPFC (fMRI-guided)
  rTMS: excitatory 5Hz. Active and Sham rTMS will be tested in a within subject design
- Active or Sham rTMS Over the Parietal Cortex (Aim1b): excitatory rTMS applied over the parietal cortex (fMRI-guided)
  rTMS: excitatory 5Hz. Active and Sham rTMS will be tested in a within subject design
- Active or Sham rTMS Over the DLPFC and the Parietal Cortex (Aim 1c); Active or Sham rTMS Over the DLPFC (Aim1a), Then Active or Sham rTMS Over the DLPFC (Aim1c): excitatory rTMS applied over the the DLPFC and the parietal cortex (fMRI-guided)
  rTMS: excitatory 5Hz. Active and Sham rTMS will be tested in a within subject design
- Total: Total of all reporting groups
Arm/Group | Active or Sham rTMS Over the DLPFC (Aim1a) | Active or Sham rTMS Over the Parietal Cortex (Aim1b) | Active or Sham rTMS Over the DLPFC and the Parietal Cortex (Aim 1c) | Active or Sham rTMS Over the DLPFC (Aim1a), Then Active or Sham rTMS Over the DLPFC (Aim1c) | Total
Number analyzed (Participants) | 83 | 42 | 58 | 1 | 184
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 57 | 18 | 58 | 1 | 134
  >=65 years | 26 | 24 | 0 | 0 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.85 (23.09) | 67.26 (6.23) | 23.65 (4.14) | 28 (1.4) | 41.31 (22.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 16 | 34 | 0 | 102
  Male | 31 | 26 | 24 | 1 | 82
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 14 | 0 | 13 | 0 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 5 | 11 | 1 | 23
  White | 62 | 37 | 33 | 0 | 132
  More than one race | 1 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 83 | 42 | 58 | 1 | 184

OUTCOME MEASURES:

1. Primary Outcome: Acute Effect of a rTMS Session on the Performance for a Working Memory Task, as Measured by Accuracy (in Percentage)
Description: Accuracy (in percentage) will be assessed to evaluate the acute effect of rTMS. The accuracy provided below are the ones obtained in the hardest condition of the working memory task.
Time Frame: During the rTMS session, on average 2 hours per visit.
Population: Subjects who completed the study. Data not collected on five subjects.
Measure: Mean (Standard Deviation); unit: percentage of accuracy
Groups:
- Active or Sham rTMS Over the DLPFC (Aim1a): excitatory rTMS applied over the DLPFC (fMRI-guided)
  rTMS: excitatory 5Hz rTMS will be used. Active and Sham rTMS will be tested in a within subject design
Arm/Group | Active or Sham rTMS Over the DLPFC (Aim1a) | Active or Sham rTMS Over the Parietal Cortex (Aim1b) | Active or Sham rTMS Over the DLPFC and the Parietal Cortex (Aim 1c)
Number analyzed (Participants) | 46 | 15 | 29
percentage of accuracy
  Active rTMS | 50.43 (7.37) | 55.42 (5.50) | 83.93 (8.09)
  Sham rTMS | 46.49 (7.35) | 57.76 (5.70) | 83.27 (10.88)

2. Primary Outcome: Acute Effect of a rTMS Session on the Performance for a Working Memory Task, as Measured by Reaction Time of Correct Response (in ms)
Description: Reaction Time of correct response (in ms) will be assessed to evaluate the acute effect of rTMS. The reaction times provided below are the ones obtained in the hardest condition of the working memory task.
Time Frame: During the rTMS session, on average 2 hours per visit
Population: Subjects who completed the study. Data not collected on five subjects.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Active or Sham rTMS Over the DLPFC (Aim1a) | Active or Sham rTMS Over the Parietal Cortex (Aim1b) | Active or Sham rTMS Over the DLPFC and the Parietal Cortex (Aim 1c)
Number analyzed (Participants) | 46 | 15 | 29
ms
  Active rTMS | 2368 (335) | 2214 (231) | 1911 (356)
  Sham rTMS | 2388 (345) | 2224 (180) | 1924 (332)

ADVERSE EVENTS:
Time Frame: During the rTMS session and a few minutes after, up to 10 minutes
Groups:
- Active rTMS Over the DLPFC (Aim1a); Sham rTMS Over the DLPFC (Aim1a): excitatory rTMS applied over the DLPFC (fMRI-guided)
  rTMS: excitatory 5Hz Active and Sham rTMS will be tested in a within subject design
- Active rTMS Over the Parietal Cortex (Aim 1b); Sham rTMS Over the Parietal Cortex (Aim 1b): excitatory rTMS applied over the parietal cortex (fMRI-guided)
  rTMS: excitatory 5Hz rTMS will be used Active and Sham rTMS will be tested in a within subject design
- Active rTMS Over the DLPFC and the Parietal Cortex (Aim 1c); Sham rTMS Over the DLPFC and the Parietal Cortex (Aim 1c); Active rTMS Over the DLPFC (Aim1a) Then Active rTMS Over the DLPFC and Parietal Cortex(Aim1c); Sham rTMS Over the DLPFC (Aim1a) Then Sham rTMS Over the DLPFC and Parietal Cortex(Aim1c): excitatory rTMS applied over the DLPFC and the parietal cortex (fMRI-guided)
  rTMS: excitatory 5Hz rTMS will be used Active and Sham rTMS will be tested in a within subject design
Arm/Group | Active rTMS Over the DLPFC (Aim1a) | Sham rTMS Over the DLPFC (Aim1a) | Active rTMS Over the Parietal Cortex (Aim 1b) | Sham rTMS Over the Parietal Cortex (Aim 1b) | Active rTMS Over the DLPFC and the Parietal Cortex (Aim 1c) | Sham rTMS Over the DLPFC and the Parietal Cortex (Aim 1c) | Active rTMS Over the DLPFC (Aim1a) Then Active rTMS Over the DLPFC and Parietal Cortex(Aim1c) | Sham rTMS Over the DLPFC (Aim1a) Then Sham rTMS Over the DLPFC and Parietal Cortex(Aim1c)
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/83 | 0/42 | 0/42 | 0/58 | 0/58 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/83 | 0/42 | 0/42 | 0/58 | 0/58 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/83 | 0/83 | 0/42 | 0/42 | 0/58 | 0/58 | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT02767323/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT02767323/SAP_001.pdf